CLINICAL TRIAL: NCT03763786
Title: A Randomised Controlled Pilot Trial of the Use of GnRH-antagonist Pituitary Suppression During Medicated Frozen-thawed Embryo Transfer (FET) Cycles
Brief Title: Frozen Embryo Transfer With GnRH-antagonist Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Collaborators: Oxford Fertility Limited, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 243105; 2018-001915-63 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2018-12-04 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No GnRH antaogonist (Experimental): Cetrorelix Acetate (NOT given) Daily 0.25mg Subcutaneous injection for 7 days
  Interventions: Drug: Cetrorelix Acetate
- Standard GnRH antoagonist (Active Comparator): Cetrorelix Acetate (control) Daily 0.25mg Subcutaneous injection for 7 days
  Interventions: Drug: Cetrorelix Acetate

INTERVENTIONS:
Drug: Cetrorelix Acetate — Used a standard
  Other Names: Cetrotide

SUMMARY:
The fertility treatment in vitro fertilisation (IVF), sometimes including intra-cytoplasmic sperm injection (ICSI), involves the creation of embryos in a laboratory. These embryos are then transferred into the womb of the patient with the hope of a resulting pregnancy and live birth. Embryos can also be cryopreserved (frozen) and stored, and then later replaced in a cycle called frozen embryo transfer (FET). There are several methods of preparing the patient's womb to receive the frozen-thawed embryo(s) but commonly embryos are replaced during a medicated cycle. Usually oestrogen and progesterone are administered to prepare the womb lining for embryo transfer at the appropriate time, and in addition a drug called a GnRH antagonist is administered to prevent a women's own hormones from interfering with this process as it is thought this might lead to higher numbers of cycles being cancelled. However, there is some suspicion that this drug (GnRH antagonist) may not be required and that women are using this drug unnecessarily.

Some clinics do not use GnRH antagonists in FET cycles, but the investigators do not know if they have higher rates of cancelled cycles as a result.

This pilot study aims to compare cycles of medicated FET using oestrogen and progesterone, either with or without pituitary suppression in the form of GnRH antagonist (Cetrotide), in patients over the next 18 months who are planning FET cycles at Oxford Fertility, UK to find out if both give the same chance of having a baby, which treatment is better for patients and to assess the feasibility of undertaking a future larger study. Cetrotide is a marketed and well-known medication and any risk or serious adverse effects are unlikely. The study is an open label prospective randomised controlled trial. Funding for the medication (Cetrotide) is provided by Oxford Fertility.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study.
* Planning to undergo medicated FET
* Blastocyst embryo in storage available for transfer

Exclusion Criteria:

* Previously randomised into the trial.
* A history of 3 or more consecutive implantation failures (after fresh or frozen embryo transfer).
* A history of recurrent miscarriage (3 or more consecutive miscarriages).
* Contraindication to the use of medications for FET cycle.
* Biopsied embryos.
* Donor embryos or eggs (use of donor sperm is not excluded).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | To treatment or pregnancy end (up to 9 months)
  Livebirth rate per FET treatment cycle

SECONDARY OUTCOMES:
Cancellation rate | Through study completion (18 months)
  Number of cycles cancelled over number of treatment cycles started

OTHER OUTCOMES:
Clinical Pregnancy Rate | To treatment or pregnancy end (up to 9 months)
  Defined as number of intrauterine pregnancies with at least one fetal heart visible on an early pregnancy ultrasound scan per treatment cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Fertility, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No